CLINICAL TRIAL: NCT03121833
Title: Randomized, Double-blind, Placebo-controlled (2: 1), Multicenter Clinical Study (IIB) for the Treatment of Stage Ⅳ Soft Tissue Sarcoma With Recombinant Human Endostatin(Endostar) Combined With Chemotherapy
Brief Title: Endostar Combined With Chemotherapy for Stage Ⅳ Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S201601-IIB
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Soft Tissue Sarcoma, Adult, Stage IIB
Keywords: Endostar; Soft Tissue Sarcoma; Chemotherapy
MeSH Terms: conditions — Sarcoma | interventions — endostar protein; Endostatins

STUDY DESIGN:
Intervention Model Description: A total of 150 cases, according to 2: 1 random into the group. Among them, 100 cases of Endostar combined chemotherapy group, 50 cases of placebo + chemotherapy group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endostar & AIM regimen / GT regimen (Experimental): Endostar & AIM regimen / GT regimen; Endostar 15mg, into 500ml 0.9% sodium chloride intravenous infusion of 3 ~ 4h, d1 ~ d14, 21-28 days for a cycle; AIM regimen is Pirarubicin (THP) + Ifosfamide (IFO), the specific dose is IFO 8-12g / m2, given 4-5 days; THP 75mg / m2, given 1-2 days; 21-28 days for a cycle; GT regimen is Docetaxel (TXT) + Gemcitabine (GEM), specific dose of Gemcitabine 1000mg / m2 (D1, D8) and Docetaxel 75mg / m2 (D8); 21-28 days for a cycle; Preferred AIM regimen, AIM regimen chemotherapy failure or can not tolerate anthracycline chemotherapy in patients with GT regimen.
  Interventions: Drug: Endostar; Drug: AIM regimen / GT regimen
- Placebo & AIM regimen / GT regimen (Placebo Comparator): Placebo + AIM regimen / GT regimen; Placebo is 500ml 0.9% sodium chloride, Intravenous 3 ~ 4h, d1 ~ d14, 21-28 days for a cycle; The chemotherapy regimen is the same as the experimental group.
  Interventions: Drug: Placebo; Drug: AIM regimen / GT regimen

INTERVENTIONS:
Drug: Endostar — Recombinant Human Endostatin Injection
  Other Names: Recombinant Human Endostatin Injection
  Arms: Endostar & AIM regimen / GT regimen
Drug: Placebo — 500ml 0.9% sodium chloride
  Other Names: Placebo(for Endostar)
  Arms: Placebo & AIM regimen / GT regimen
Drug: AIM regimen / GT regimen — "Pirarubicin (THP) + Ifosfamide (IFO)" / "Docetaxel (TXT) + Gemcitabine (GEM)"

SUMMARY:
This is a randomized, double-blind, placebo-controlled (2: 1), multicenter clinical phase II clinical trial evaluating the efficacy and safety of Endostar combined with chemotherapy for stage IV soft tissue sarcoma.

DETAILED DESCRIPTION:
The prognosis of sarcoma patients in stage IV is poor. For STS, the response rate of chemotherapy is only 20-35% and the median survival time is about 12 months. The 5 year survival rate is lower than 10% reported in several large-scale studies. Although chemotherapy plays a major role in the treatment of advanced STS, the classic chemotherapy agents are not curative. Combination chemotherapy or dose-dense regimens have largely failed to improve the response rates. Long-term using of cytotoxic drugs increased the risk of toxicity in patients. Endostatin is the strongest endogenous angiogenesis inhibitor, which inhibits vascular endothelial growth factor (VEGF) expression and then inhibits tumor angiogenesis . Endostar, is a novel recombinant human endostatin, with advantages of long half-life, stable and low cost. Recently, a study of Endostar combined with chemotherapy in the treatment of advanced soft tissue sarcoma indicated resulted in a higher clinical benefit response (CBR) and longer progression-free survival (PFS), with tolerable side effects. However this study included the patients with stage IIB-IV soft tissue sarcomas and did not include specific pathologic information. Thus this clinical trial is designed to compare the efficacy and safety of endostar combined with chemotherapy versus chemotherapy alone in stage IV patients with soft tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered to participate in this study, signed informed consent;
* Pathological diagnosis of stage Ⅳ of soft tissue sarcoma patients, clinical staging using the American Cancer Research Joint Commission (AJCC) TNM staging criteria. There is at least one extracranial measurable lesion based on CT or MRI.
* 18 to 75 years old; the patient's physical condition Karnofsky score ≧ 60 points; ECG, blood, liver and kidney function were no abnormalities; expected survival ≧ 6 months.
* Major organ function within 7 days prior to treatment, meeting the following criteria:

  1. Blood routine examination criteria (14 days without blood transfusion):

     * ①hemoglobin (HB) ≥ 90g / L;② neutrophil absolute value (ANC) ≥ 1.5 × 109 / L;③ platelet (PLT) ≥ 80 × 109 / L.
  2. Biochemical tests to meet the following criteria:

     * ①Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);② Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5 × ULN, such as liver metastasis, the ALT and AST ≤ 5×ULN;③ Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 60ml / min;
  3. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ normal low (50%).
* Women of childbearing age should agree that contraceptive measures (such as intrauterine devices, birth control pills or condoms) must be used within the study period and within 6 months after the end of the study; the serum or urine pregnancy test is negative within 7 days prior to the study For non-lactating patients; men should agree to patients who have contraindications during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Patients who had previously used Endostar injections;
* Patients who have received antiangiogenic therapy or other targeted treatment for no more than 3 months, such as Endostar, Erlotinib, Sunitinib, Sorafenib, Avastin, Imatinib, Famitinib, Pazopanib and other drugs.
* 5 years or present at the same time suffering from other malignant tumors. Cured cervix in situ cancer, non-melanoma skin cancer and superficial bladder tumors except. [Ta (non-invasive tumor), Tis (orthotopic carcinoma) and T1 (tumor infiltrating basement membrane)];
* During the first 4 weeks of the group or during the study period, systemic anti-tumor therapy was planned, including cytotoxic therapy and immunotherapy. Intravenous radiotherapy (EF-RT) was performed 4 weeks prior to grouping or restricted radiotherapy was performed within 2 weeks prior to grouping to assess tumor lesions;
* Due to any previous treatment caused by the CTC AE (4.0) level 1 or more of the mitigated toxicity, excluding hair loss;
* Patients with symptoms or symptoms of control less than 2 months of brain metastases;
* Any patient with severe and / or uncontrolled disease, including:

  1. Patients with poor blood pressure control. (Systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg);
  2. Myocardial ischemia or myocardial infarction, arrhythmia (including QTC ≥480 ms) and ≥ 2 levels of congestive heart failure (NYHA classification)
  3. Active or uncontrollable serious infections (≥CTC AE Level 2 infection);
  4. Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis to be treated with antiretroviral therapy;
  5. Renal failure requires hemodialysis or peritoneal dialysis;
  6. History of immunodeficiency, including HIV positive or other acquired, congenital immune deficiency disease, or a history of organ transplantation;
  7. Poor control of diabetes (fasting blood glucose (FBG)> 10mmol / L);
  8. Urine Urine Urine protein ≥ ++, and confirmed 24 hours urine protein> 1.0 g;
  9. Patients with a seizure and need treatment.
* Significant surgical treatment, biopsy or traumatic injury was received within 28 days prior to the grouping;
* Regardless of the severity of the presence of any signs of bleeding or medical history of patients; in the first 4 weeks before the group, any bleeding or bleeding events ≥ CTCAE3 patients, there is no healing wounds, ulcers or fractures;
* Subluxation / venous thrombosis events occurred within 6 months before the group, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
* Have a history of psychiatric abuse and can not quit or have mental disorders;
* Four weeks before the group participated in other clinical trials of anti-tumor drugs;
* According to the researcher's judgment, there are other comorbidities that seriously endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 year
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Disease control rate(DCR） | 2 year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）

OTHER OUTCOMES:
Objective tumor response rate(ORR) | 2 year
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
Overall survival(OS) | 3 year
  OS is defined as the length of time from random assignment to death or to last contact.
Adverse Events(AEs) | 2 year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jilong Yang, M.D., Ph.D., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Hospital & Institute, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No